CLINICAL TRIAL: NCT05247216
Title: A Multicenter, Randomized, Double-blind Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Hemay007 in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Phase 2 Study of Hemay007 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM007RA2S01; CTR20201916 (Other: Center for Drug Evaluation, NMPA)
Record Dates: First submitted 2021-05-31; First posted 2022-02-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate to severe Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hemay007 800 mg QD group (Experimental): Drug: 800mg QD of Hemay007; daily oral administrtion for 12 weeks
  Interventions: Drug: Hemay007 800 mg QD group
- Hemay007 1200 mg QD group (Experimental): Drug: 1200mg QD of Hemay007; daily oral administrtion for 12 weeks
  Interventions: Drug: Hemay007 1200 mg QD group
- Hemay007 600 mg QD group (Experimental): Drug: 600mg QD of Hemay007; daily oral administrtion for 12 weeks
  Interventions: Drug: Hemay007 600 mg QD group
- placebo group (Placebo Comparator): Drug: placebo of Hemay007; daily oral administrtion for 12 weeks
  Interventions: Drug: Hemay007 placebo group

INTERVENTIONS:
Drug: Hemay007 800 mg QD group — daily oral administrtion of Hemay007 800 mg QD for 12 weeks, 4 tablets of 200mg Hemay007 and 2 tablets of placebo.
  Arms: Hemay007 800 mg QD group
Drug: Hemay007 1200 mg QD group — daily oral administrtion of Hemay007 1200 mg QD for 12 weeks, 6 tablets of 200mg Hemay007.
  Arms: Hemay007 1200 mg QD group
Drug: Hemay007 600 mg QD group — daily oral administrtion of Hemay007 600 mg QD for 12 weeks, 3 tablets of 200mg Hemay007 and 3 tablets of placebo.
  Arms: Hemay007 600 mg QD group
Drug: Hemay007 placebo group — daily oral administrtion of placebo for 12 weeks 6 tablets of placebo.
  Arms: placebo group

SUMMARY:
This is a multicenter, randomized, double-blind phase2 study to evaluate the safety and investigate the efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of Hemay007 in Patients with moderate to severe Rheumatoid Arthritis who are on a stable dose of DMARDs.

DETAILED DESCRIPTION:
This study adopts a multi-center, randomized, double-blind clinical study design. Patients with moderate to severe active rheumatoid arthritis who meet the inclusion criteria but do not meet the exclusion criteria will be randomly assigned into the 600 mg QD group, 800 mg QD group, 1200 mg QD group and placebo group at a ratio of 1:1:1:1, with about 35 subjects in each group. Patients in all the groups will be treated with Hemay007 or placebo for 12 weeks, and observed for 4 weeks after the treatment. This study is to evaluate the safety and investigate the efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of Hemay007 in Patients with moderate to severe Rheumatoid Arthritis who are on a stable dose of DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old (both ends included, subject to the date of signing the informed consent form), male or female.
* According to the 1987 American College of Rheumatology (ACR) or 2010 ACR/EULAR classification diagnostic criteria, the diagnosis was rheumatoid arthritis, and the course of disease was ≥12 weeks.
* If rheumatoid arthritis is moderately or severely active, the disease activity during the screening period and the baseline period must meet the following criteria:

Swollen joints count (SJC) ≥ 6 (based on 66 joint count) and tender joints count (Tender joints count: TJC) ≥ 6 (based on 68 joint count) (if the same joint has both swelling and Tenderness, this joint is included in the counts of swollen joints and tender joints). Joints that have undergone major surgery and joints that have been intraarticularly injected with corticosteroids or hyaluronic acid within 2 weeks before screening or 6 weeks before randomization are not counted in TJC (tender joint count) and SJC (swollen joint count) count.

Erythrocyte sedimentation rate (ESR)>28mm/h or C-reactive protein (CRP) (or hypersensitive CRP (hsCRP))>1.5 times the upper limit of the normal range (ULN).

* Subjects who have used at least one rheumatism-improving drug (DMARDs) treatment, but have poor efficacy (drug time ≥12 weeks, DAS28>3.2) or intolerance (drug use interrupted due to adverse reactions) By.
* Methotrexate (MTX, 7.5-25 mg/week) has been used continuously for at least 12 weeks, and the dose has been stabilized for at least 4 weeks before the first administration, and a stable medication regimen shall be maintained during the trial period.
* If the subject is taking non-steroidal anti-inflammatory drugs (NSAIDS≤1), the dose must be stabilized for at least 2 weeks before the first administration. And/or oral corticosteroids (prednisone ≤10mg/day or equivalent dose), the dose must have been stabilized for at least 4 weeks before the first dose, and a stable medication regimen should be maintained during the trial period.
* The time to stop medication before the first dose meets the following criteria:

For traditional medicines for improving rheumatism, such as:Sulfasalazine, hydroxychloroquine, cyclosporine, azathioprine drugs: stop the drug for 4 weeks before the first administration;

Leflunomide: The drug should be stopped for 12 weeks before the first dose, or cholestyramine should be eluted for 11 days, and the drug should be stopped for 7 days before the first dose.

Cyclophosphamide: Stop the drug for 8 weeks before the first dose.

For biological agents, such as: Anakinra, Etanercept: Stop the drug for 4 weeks before the first dose; Adalimumab: stop the drug for 6 weeks before the first dose;Infliximab, golimumab: stop the drug for 8 weeks before the first administration; Certuzumab: stop the drug for 10 weeks before the first dose; Tocilizumab, abatizumab: stop the drug for 12 weeks before the first administration; Cell depletion therapy, such as rituximab: stop the drug for 1 year before the first dose.

Others, such as: JAK inhibitors, such as tofacitinib, need to be stopped for 1 year before the first dose; Iguratimod: need to stop the drug for 4 weeks before the first dose; Intra-articular, intramuscular or intravenous injection of steroids: stop the drug for 4 weeks before the first dose; Plasma exchange: stop for 12 weeks before the first dose; Chinese medicine, Chinese patent medicine and Chinese medicine single medicine treatment (including tripterygium wilfordii, total glucosides of paeony, sinomenine): stop the medicine for 2 weeks before the first administration;Any other drugs not mentioned: The drug should be stopped for 4 weeks or more than 5 half-lives before the first administration, whichever is longer.

* Take medically approved non-drug contraceptive measures (such as drug-free intrauterine devices, condoms, female sterilization, and male sterilization) during the entire trial period and at least 3 months after the end of the medication, and no Pregnancy planner.
* Those who understand, voluntarily sign the informed consent form, and comply with the requirements of the research plan.

Exclusion Criteria:

* Those who are known to be allergic to any component of hemay007 tablets.
* Those who have received any medical supportive treatments (such as whitening drugs, drugs for anemia (except folic acid), liver-protecting and enzyme-lowering drugs, blood transfusions, etc.) within 2 weeks before screening.
* The joint function classification of rheumatoid arthritis is Grade IV or those who need to stay in bed/sedentary wheelchair for a long time due to limited joint function activities.
* Those who have taken gold preparations or penicillamine in the past or during screening.
* In the past or at the time of screening, there were other inflammatory joint diseases other than RA (such as: gout, reactive arthritis, psoriatic arthritis, spondyloarthropathy, etc.). Or other joint diseases that may affect the evaluation of curative effect (such as: osteoarthritis with obvious joint pain), the investigator judged that it is not suitable to join the trial.
* Past or at the screening systemic autoimmune diseases (such as systemic lupus erythematosus, Felty syndrome, scleroderma, primary Sjogren's syndrome, etc., except for secondary Sjogren's syndrome), or organ-specific For autoimmune diseases (such as hyperthyroidism, Hashimoto's thyroiditis, etc.), the investigator has judged that it is not suitable to join this trial.
* Patients with acute myocardial infarction, unstable angina pectoris, stroke, and cardiac insufficiency (New York Heart Association (NYHA) cardiac function classification III/IV) within 6 months before screening.
* The cardiovascular, liver, kidney, lung, digestive tract, nervous system and other serious diseases (such as: poorly controlled severe diabetes, hypertension, interstitial pneumonia, obstructive Lung disease, bronchospasm, etc.), the investigator judged that it is not suitable to join the research.
* At the time of screening, the laboratory test (γ-interferon release test) was positive and met any of the following conditions. The investigator judged that the tuberculosis infection or suspected infection was.

Chest imaging examination showed suspected tuberculosis infection; Active pulmonary tuberculosis; Those who have had active Mycobacterium tuberculosis infection within 3 years before screening; People who have been in contact with or have active tuberculosis in the home environment.

* Active infection (virus, bacteria, fungus, parasite infection) during screening, mild fungal infection (such as mild nail infection), or severe infection within 6 months before screening, as judged by the investigator Those who are not suitable to join this trial.
* Patients with any type of malignant tumor in the past or at the time of screening.
* Patients who have demyelinating diseases of the central nervous system (such as multiple sclerosis, optic neuritis, etc.) in the past or during screening, or have neurological symptoms suggestive of demyelinating diseases.
* Those who have suffered severe trauma, fracture or joint surgery within 4 weeks before screening, or are expected to undergo major surgery during the trial period.
* Those who have undergone surgery that may affect drug absorption, distribution, metabolism, and excretion within 3 months before screening, or are expected to undergo such surgery during the trial period.
* The laboratory examination meets any of the following conditions, and the investigator judges that it is not suitable to participate in this trial:

Renal function: blood creatinine>1.5×ULN;

Liver function: ALT or AST>1.5×ULN, or TBIL>1.5×ULN;

Blood routine: white blood cell count (WBC) <3.0×10^9/L, absolute neutrophil count (ANC) <1.5×10^9/L, absolute lymphocyte count (ALC) <0.5×10^9/L, platelet count (PLT) )<100×10^9/L, hemoglobin (HGB)<85g/L;

Blood biochemistry: triglyceride>10mmol/L.

* Those who have a history of smoking, alcoholism, or drug abuse within 12 months before screening.
* Active hepatitis B (hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA higher than the local normal test value), hepatitis C, or syphilis infection during screening.
* People with other primary or secondary immunodeficiencies in the past or at the time of screening, including patients with a history of HIV infection and positive HIV test results.
* Those who have participated in other clinical studies within 3 months before screening.
* Women who are preparing for pregnancy, pregnancy, lactation, or who become pregnant during the planned trial period.
* The investigator believes that it is not suitable to participate in this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
ACR20 | week 4
  The proportion of subjects who achieved ACR 20 remission at the week 4.
ACR20 | week 8
  The proportion of subjects who achieved ACR 20 remission at the week 8.
ACR20 | week 12
  The proportion of subjects who achieved ACR 20 remission at the week 12.
ACR20 | week 16
  The proportion of subjects who achieved ACR 20 remission at the week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, M.D., Principal Investigator — Southern Hospital of Southern Medical University
Locations (41):
- China (41):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University The Sixth Affiliated Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Hebei PetroChina Central Hospital, Langfang, Hebei
  - Henan University of Science and Technology The First Affiliated Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Loudi Central Hospital, Loudi, Hunan
  - The First Affiliated Hospital of Shaoyang University, Shaoyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First People's Hospital of Jiujiang City, Jiujiang, Jiangxi
  - Nanchang University The Second Affiliated Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang City People's Hospital, Pingxiang, Jiangxi
  - Jilin University Sino-Japanese Friendship Hospital, Changchun, Jilin
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Panjin Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Ningxia Hui Autonomous Region People's Hospital, Yinchuan, Ningxia
  - Heze Municipal Hospital, Heze, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Yantai Mountain Hospital, Yantai City, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Shanghai University of Traditional Chinese Medicine Affiliated Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Changzhi Medical College Peace Hospital, Changzhi, Shanxi
  - Jinzhong First People's Hospital, Jinzhong, Shanxi
  - Guangyuan Central Hospital, Guangyuan, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Huzhou Third People's Hospital, Huzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Beijing Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
It is yet decided not to share the individual participant data (IPD) to other researchers.